CLINICAL TRIAL: NCT03254069
Title: Changes in Occlusal Bite Force Following Placement of Stainless Steel Crowns on Primary Molars in Children
Brief Title: Occlusal Bite Force Changes After Placement of Stainless Steel Crowns in Children
Acronym: OBF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Principal Investigator, Arwa Issa Owais, Principal Investigator, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Occlusal Bite Force
Record Dates: First submitted 2016-04-08; First posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stainless Steel Crown Arm (Experimental): Children with SSCs placed and followed longitudinal. Consent was obtained from all parents and verbal assent was obtained. The following data was collected: Demographic Data of the Children, clinical examination, radiographs, treatment planning, details of stainless steel crowns placement, OBF measurements were made before the SSC placement and periodically post placement
  Interventions: Device: Stainless Steel Crowns
- Control Arm (No Intervention): A second group consisted of twenty-two children (11 females and 11 males; a mean age of 5.20 ± 0.36 years) were selected to act as a control sample and received no dental treatment. MOBF was recorded in these subjects at T0 and T5 (6 months after).

INTERVENTIONS:
Device: Stainless Steel Crowns — SSCs were placed on children's primary molars, and bite force was registered prior to the study, and periodically after the study.
  Other Names: SSCs
  Arms: Stainless Steel Crown Arm

SUMMARY:
The aim of this study was to determine if restoring primary molars with SSCs would improve children's OBF.

DETAILED DESCRIPTION:
Occlusal bite force (OBF) is an indicator of the functional status of the masticatory system. The level of maximum occlusal bite force (MOBF) results from the combined action of the jaw elevator muscles modified by jaw biomechanics and reflex mechanisms. The measurement of OBF has been widely used in dentistry to provide useful data for the evaluation of jaw muscle function and activity as well as effectiveness of prosthetic therapy.

Many indicators have been believed to assess the functional status of the masticatory system, such as body size, bite force, number of functional tooth units, and the occlusal contact area. Dental status formed with dental fillings, dentures, position and the number of teeth is an important factor in the value of the OBF.

Many studies were conducted to evaluate the effect of dental caries on OBF. Tsai et al. found a negative correlation between MOBF and the number of decayed teeth. Su et al. reported that the overall tooth decay was not related to the strength of OBF. They suggested that the severity of tooth decay may be more important than the number of teeth exhibiting decay.

Stainless Steel Crowns (SSCs) are considered the treatment of choice for severely decayed but restorable primary molars. A recent systematic review by Seale and Randall confirmed their previous work and reviews and appeared to continue to be supportive and in favor of SSCs.

SSCs has been blamed for premature contact related discomfort in the first few weeks after placement of SSCs. Zee and Amerongen reported that premature contacting SSC restored teeth will equilibrate over time and return to pretreatment levels in 15 to 30 days.

Several opinions have been reported by parents, children and dentists regarding the improved mastication efficiency after placement of the SSCs. However, the effects of SSCs placement on primary molars on OBF have not yet been investigated

ELIGIBILITY:
Inclusion Criteria:- Caucasian

* Healthy child
* In the primary dentition stage
* Class I occlusion
* No facial asymmetry
* No cross bite
* Have caries in the eight primary molars indicating placement of SSCs, with no reported pain on biting and no previous restorations
* No gingival inflammation
* No para functional habits

Exclusion Criteria: did not meet the inclusion criteria stated above

-

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum Occlusal Bite Force (MOBF) | Six Months post placement
  Occlusal Bite Force will be measured in Newton

CONTACTS AND LOCATIONS:
Overall Officials: arwa Owais, BDS, Principal Investigator — Jordan University of Science & Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mountain G, Wood D, Toumba J. Bite force measurement in children with primary dentition. Int J Paediatr Dent. 2011 Mar;21(2):112-8. doi: 10.1111/j.1365-263X.2010.01098.x. Epub 2010 Aug 20. PMID 20731734
- [Result] Koc D, Dogan A, Bek B. Bite force and influential factors on bite force measurements: a literature review. Eur J Dent. 2010 Apr;4(2):223-32. PMID 20396457
- [Result] Ohira A, Ono Y, Yano N, Takagi Y. The effect of chewing exercise in preschool children on maximum bite force and masticatory performance. Int J Paediatr Dent. 2012 Mar;22(2):146-53. doi: 10.1111/j.1365-263X.2011.01162.x. Epub 2011 Jul 22. PMID 21781200
- [Result] Owens S, Buschang PH, Throckmorton GS, Palmer L, English J. Masticatory performance and areas of occlusal contact and near contact in subjects with normal occlusion and malocclusion. Am J Orthod Dentofacial Orthop. 2002 Jun;121(6):602-9. doi: 10.1067/mod.2002.122829. PMID 12080313
- [Result] Oueis H. Factors affecting masticatory performance of Japanese children. Int J Paediatr Dent. 2009 May;19(3):201-5. doi: 10.1111/j.1365-263X.2008.00965.x. Epub 2009 Jan 16. PMID 19207738
- [Result] Tsai HH. Maximum bite force and related dental status in children with deciduous dentition. J Clin Pediatr Dent. 2004 Winter;28(2):139-42. doi: 10.17796/jcpd.28.2.j42870t47q4n1715. PMID 14969373
- [Result] Seale NS. Stainless steel crowns improve success rate of root canal treatment in primary teeth. J Evid Based Dent Pract. 2005 Dec;5(4):205-6. doi: 10.1016/j.jebdp.2005.09.011. No abstract available. PMID 17138373
- [Result] Atieh M. Stainless steel crown versus modified open-sandwich restorations for primary molars: a 2-year randomized clinical trial. Int J Paediatr Dent. 2008 Sep;18(5):325-32. doi: 10.1111/j.1365-263X.2007.00900.x. Epub 2008 Mar 6. PMID 18328050
- [Result] Seale NS, Randall R. The use of stainless steel crowns: a systematic literature review. Pediatr Dent. 2015 Mar-Apr;37(2):145-60. PMID 25905656
- [Result] van der Zee V, van Amerongen WE. Short communication: Influence of preformed metal crowns (Hall technique) on the occlusal vertical dimension in the primary dentition. Eur Arch Paediatr Dent. 2010 Oct;11(5):225-7. doi: 10.1007/BF03262751. PMID 20932395
- [Result] Kindelan SA, Day P, Nichol R, Willmott N, Fayle SA; British Society of Paediatric Dentistry. UK National Clinical Guidelines in Paediatric Dentistry: stainless steel preformed crowns for primary molars. Int J Paediatr Dent. 2008 Nov;18 Suppl 1:20-8. doi: 10.1111/j.1365-263X.2008.00935.x. PMID 18808544
- [Result] Owais AI, Shaweesh M, Abu Alhaija ES. Maximum occusal bite force for children in different dentition stages. Eur J Orthod. 2013 Aug;35(4):427-33. doi: 10.1093/ejo/cjs021. Epub 2012 Apr 19. PMID 22518063
- [Result] Serra MD, Gambareli FR, Gaviao MB. A 1-year intraindividual evaluation of maximum bite force in children wearing a removable partial dental prosthesis. J Dent Child (Chic). 2007 Sep-Dec;74(3):171-6. PMID 18482509